CLINICAL TRIAL: NCT05764369
Title: Optimizing Residential Treatment Gains for Adolescents Through Tailored Behavioral Parent Training
Brief Title: Optimizing Residential Treatment Gains for Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Kayla Herbell, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022B0315
Record Dates: First submitted 2023-02-13; First posted 2023-03-10 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Parenting; Adolescent - Emotional Problem; Mental Disorder in Adolescence

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will not know which group they are assigned to, however, study staff will know.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Parenting Wisely Residential Treatment (PWRT) (Experimental): In the PWRT condition, parents will complete a total of ten web-based modules in an online parent training program called Parenting Wisely. Each week, parents will also attend a 90-minute facilitated discussion group via Zoom. Parents will complete assessments at baseline (T1), six weeks post-baseline (T2), and six months post-baseline (T3) via REDCap. While adolescents (n=60) will not directly receive the intervention, they will complete assessments at baseline, six weeks post-baseline (T2), and six months post-baseline (T3).
  Interventions: Behavioral: Parenting Wisely Residential Treatment (PWRT)
- Treatment as Usual (TAU) (Placebo Comparator): The TAU condition is the standard of care offered to parents in RT settings. Parents in the TAU condition will receive traditional programming, including family therapy offered weekly during the RT admission. Parents will attend discharge planning meetings with caseworkers (if assigned) to discuss the adolescent's progress, continued treatment needs, safety plans, upcoming appointments, and medication needs. Following discharge, programs frequently recommend follow-up with an outpatient provider for medication management and therapy for the adolescent. Parents will complete assessments at baseline (T1), six weeks post-baseline (T2), and six months post-baseline (T3) via REDCap. While adolescents (n=60) will not directly receive the intervention, they will complete assessments at baseline, six weeks post-baseline (T2), and six months post-baseline (T3).
  Interventions: Behavioral: TAU

INTERVENTIONS:
Behavioral: Parenting Wisely Residential Treatment (PWRT) — PWRT experimental intervention
  Other Names: Parenting Wisely; PW
  Arms: Parenting Wisely Residential Treatment (PWRT)
Behavioral: TAU — The TAU condition is the standard of care offered to parents in RT settings.
  Arms: Treatment as Usual (TAU)

SUMMARY:
The goal of this randomized controlled trial is to determine the feasibility, acceptability, and preliminary effects of a web-based parent training augmented with facilitated parent groups. This hybrid group-based parenting program (called Parenting Wisely for Residential Treatment; PWRT) is designed to prepare parents for the reintegration of their adolescents in the home after intensive psychiatric residential treatment. Researchers will compare PWRT to treatment as usual to determine whether PWRT effects target mechanisms (i.e., family function, social support, parental self-efficacy, parenting practices) and adolescent outcomes (i.e., internalizing and externalizing behaviors, placement restrictiveness).

DETAILED DESCRIPTION:
A randomized controlled trial (RCT) design is employed to evaluate the feasibility, acceptability, engagement of target mechanisms, and preliminary effects of PWRT in parents with adolescents transitioning from residential treatment (RT) to the community. Parents (n=60) will be randomly assigned to receive Parenting Wisely augmented with facilitated discussion groups (referred to as PWRT; n=30) or treatment-as-usual (TAU; n=30). In the PWRT condition, parents will complete 2 web-based modules in an online parent training program called Parenting Wisely. Parents will also attend a 90-minute discussion group via Zoom. The RCT will allow for testing of target mechanism engagement (i.e., parental self-efficacy, parenting behaviors, social support, family function) and the intervention's effects on adolescent outcomes (i.e., internalizing behaviors, externalizing behaviors, placement restrictiveness). Parents will complete assessments at baseline (T1), six weeks post-baseline (T2), and six months post-baseline (T3) via REDCap. While adolescents (n=60) will not directly receive the intervention, they will complete assessments at baseline, six weeks post-baseline (T2), and six months post-baseline (T3).

Aim 1: Evaluate the feasibility and acceptability of PWRT. 1a. Evaluate the feasibility of PWRT by tracking the frequency, dose, and duration. 1b. Evaluate the acceptability of PWRT for parents with adolescents in RT.

Aim 2: Determine the effects of PWRT on the target mechanisms compared to the TAU condition from baseline to 6-weeks and 6-months post-baseline.

Aim 3: Determine the effects of PWRT on adolescent outcomes compared to the TAU condition from baseline to 6-weeks and 6-months post-baseline. 3a. Determine if changes in the target mechanisms are associated with adolescent outcomes at six weeks and six months post-baseline.

Exploratory Aim: Explore the feasibility of collecting data from adolescents in an RT facility by tracking frequency (recruitment, enrollment, retention rates), duration (time between parent consent and assent; survey duration), and barriers to data collection.

ELIGIBILITY:
Parent Inclusion Criteria:

* Caregiver (e.g., biological, step, kin, foster, adoptive) to an adolescent aged 11-17 years old admitted to psychiatric residential treatment;
* The caregiver is allowed contact with the adolescent;
* Has access to a device (e.g., smartphone) with internet access.

Adolescent Inclusion Criteria:

* Ability to understand and willingness to provide written assent
* Legal guardian provides written consent;
* Currently or previously admitted to psychiatric residential treatment
* Aged 11-17 years at enrollment;

Parent and Adolescent Exclusion Criteria:

- Not able to speak English

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-08-31 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-06-02 (Actual)

PRIMARY OUTCOMES:
Group Attendance (Feasibility) | Mean calculated at 6-weeks post-baseline
  The mean number of groups attended by participants.
Module Completion (Feasibility) | Mean calculated at 6-weeks post-baseline
  The mean number of modules completed by participants in Parenting Wisely.
Module Duration (Feasibility) | Mean calculated at 6-weeks post-baseline
  The mean time participants spent completing one module in Parenting Wisely.
Group Duration (Feasibility) | Mean calculated at 6-weeks post-baseline
  The mean amount of time participants spent in a single session of the group.
PWRT Acceptability | Mean calculated at 6-weeks post-baseline
  Participants will complete a satisfaction survey to evaluate the acceptability of PWRT. The satisfaction survey consists of 13-items. Total scores range from 0-39; higher scores indicate greater perceptions of acceptability.

SECONDARY OUTCOMES:
Change in Adolescent Internalizing Behaviors | Change from baseline to 6-months post-baseline
  Adolescent internalizing behaviors will be assessed using the Brief Problem Monitor (BPM) for ages 6 to 18. The BPM consists of 19 items derived from the Child Behavior Checklist. The subscales include internalizing, externalizing, and attention subscales. Raw scores range from 0-38; higher scores indicate greater internalizing behaviors.
Change in Adolescent Internalizing Behaviors | Change from baseline to 6-weeks post-baseline
  Adolescent internalizing behaviors will be assessed using the Brief Problem Monitor (BPM) for ages 6 to 18. The BPM consists of 19 items derived from the Child Behavior Checklist. The subscales include internalizing, externalizing, and attention subscales. Raw scores range from 0-38; higher scores indicate greater internalizing behaviors.
Change in Adolescent Externalizing Behaviors | Change from baseline to 6-weeks post-baseline
  Adolescent externalizing behaviors will be assessed using the Brief Problem Monitor (BPM) for ages 6 to 18. The BPM consists of 19 items derived from the Child Behavior Checklist. The subscales include internalizing, externalizing, and attention subscales. Raw scores range from 0-38; higher scores indicate greater externalizing behaviors.
Change in Adolescent Externalizing Behaviors | Change from baseline to 6-months post-baseline
  Adolescent externalizing behaviors will be assessed using the Brief Problem Monitor (BPM) for ages 6 to 18. The BPM consists of 19 items derived from the Child Behavior Checklist. The subscales include internalizing, externalizing, and attention subscales. Raw scores range from 0-38; higher scores indicate greater externalizing behaviors.
Change in Restrictiveness of Living Environment | Change from baseline to 6-weeks post-baseline
  The Restrictiveness Evaluation Measure (REM) will be administered to evaluate perceptions of adolescent placement restrictiveness. The REM was designed and tested in residential treatment settings. There are two subscales; one scale identifies 25 placement settings varying in restrictiveness and the second subscale consists of questions about the activity and lifestyle restrictions in such placements. Total scores range from 24-120; higher scores indicate more restrictive living environments.
Change in Restrictiveness of Living Environment | Change from baseline to 6-months post-baseline
  The Restrictiveness Evaluation Measure (REM) will be administered to parents and adolescents to evaluate perceptions of adolescent placement restrictiveness. The REM was designed and tested in residential treatment settings. There are two subscales; one scale identifies 25 placement settings varying in restrictiveness and the second subscale consists of questions about the activity and lifestyle restrictions in such placements. Total scores range from 24-120; higher scores indicate more restrictive living environments.
Change in Family Function | Change from baseline to 6-weeks post-baseline
  The McMaster Family Assessment Device (FAD) will be administered to parents to evaluate changes in family function. The FAD consists of 60-items that assess seven domains of family function: problem-solving, family roles, communication, affective involvement, affective responsiveness, behavioral control, general functioning. Total scores range from 60-240; higher scores indicate better family function.
Change in Family Function | Change from baseline to 6-months post-baseline
  The McMaster Family Assessment Device (FAD) will be administered to parents to evaluate changes in family function. The FAD consists of 60-items that assess seven domains of family function: problem-solving, family roles, communication, affective involvement, affective responsiveness, behavioral control, general functioning. Total scores range from 60-240; higher scores indicate better family function.
Change in Social Support | Change from baseline to 6-weeks post-baseline
  The Medical Outcomes Study (MOS) Social Support Survey will be administered to parents to evaluate changes in social support. The MOS consists of 19-items that assess five social support domains: emotional support, informational support, tangible support, affectionate support, and positive social interaction. Total scores range from 20-100; higher scores indicate greater social support.
Change in Social Support | Change from baseline to 6-months post-baseline
  The Medical Outcomes Study (MOS) Social Support Survey will be administered to parents to evaluate changes in social support. The MOS consists of 19-items that assess five social support domains: emotional support, informational support, tangible support, affectionate support, and positive social interaction.Total scores range from 20-100; higher scores indicate greater social support.
Change in Parenting Self Efficacy | Change from baseline to 6-weeks post-baseline
  Parents will complete the Parenting Sense of Competence Scale (PSOC) to evaluate changes in parental self-efficacy. The PSOC consists of 17-items and is designed for parents with children aged birth to 17. The two subscales in the PSOC are satisfaction and efficacy. Total scores range from 17-102; higher scores indicate greater perceptions of self-efficacy and confidence.
Change in Parenting Self Efficacy | Change from baseline to 6-months post-baseline
  Parents will complete the Parenting Sense of Competence Scale (PSOC) to evaluate changes in parental self-efficacy. The PSOC consists of 17-items and is designed for parents with children aged birth to 17. The two subscales in the PSOC are satisfaction and efficacy. Total scores range from 17-102; higher scores indicate greater perceptions of self-efficacy and confidence.

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio State University College of Nursing, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from this study will be submitted to the National Institute of Mental Health Data Archive (NDA) at the National Institutes of Health (NIH). If a participant consents to having their data deposited in the NDA, the study team will create a global unique identifier (GUID) using the NDA GUID Tool. The GUID Tool requires a participant's full name, birth date, city of birth, and sex at birth to generate an alphanumeric code that is used to identify a participant across studies. In this study, data that will be deposited will include primary outcomes measures such as The Brief Problem Monitor, the Restrictiveness Evaluation Measure, Parenting Sense of Competence Scale, Adult-Adolescent Parenting Inventory, Medical Outcomes Study Social Support Survey, and McMaster Family Assessment Device. See NDA for more details.
Supporting Information: Study Protocol, ICF
Time Frame: Raw experimental data (both baseline and longitudinal) will not be released/shared until publication or 12 months after the project end date, whichever comes first.
Access Criteria: The NIH will provide access to scientific investigators for research purposes. Qualified researchers who have completed a Data Use Certification and received approval from the NDA Data Access Committee (DAC) may be approved to access broadly shared data. A separate request process exists for access to data in federated sources. Additionally, the DAC and support staff at NIH have access to NDA shared data.

REFERENCES:
- [Derived] Herbell K, Breitenstein SM, Tan A, Melnyk BM, Thai AT, Berger S. Families in transition (FIT) study protocol: feasibility, acceptability and preliminary effects of a group-based parent training in parents of youth in psychiatric residential treatment. BMJ Open. 2024 May 30;14(5):e080603. doi: 10.1136/bmjopen-2023-080603. PMID 38816058